CLINICAL TRIAL: NCT07141186
Title: A Prospective, Single-Arm, Phase II Trial of QL1706 in Patients With Recurrent and/or Metastatic Cervical Cancer Who Had Developed Resistance to Prior PD-1/PD-L1 Antibody Therapy
Brief Title: QL1706 in Patients With Recurrent and Metastatic Cervical Cancer Resistant to Prior PD-1/PD-L1 Antibody Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Zhiyong Yuan, Head of Radiotherapy Department, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020250707083952035
Record Dates: First submitted 2025-07-23; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Cervical Cancer; Cervical Cancer Metastatic; Cervical Cancer Recurrent; Cervical Adenocarcinoma; Cervical Cancer Squamous Cell
Keywords: cervical cancer; immunotherapy; PD-1/CTLA-4 bispecific antibody; QL1706; PD-1 resistant
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1/CTLA-4 bispecific antibody treatment group (Experimental): Enrolled patients will receive intravenous infusion of QL1706 once every 3 weeks at a dose of 5.0 mg/kg until disease progression, death, intolerable treatment toxicity, or withdrawal from the clinical trial for any reason.
  Interventions: Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4)

INTERVENTIONS:
Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4) — Enrolled patients will receive intravenous infusion of QL1706 once every 3 weeks at a dose of 5.0 mg/kg until disease progression, death, intolerable treatment toxicity, or withdrawal from the clinical trial for any reason.

SUMMARY:
To explore the efficacy and safety of administrating QL1706 in patients with recurrent and/or metastatic cervical cancer who had developed resistance to prior PD-1/PD-L1 antibody therapies.

DETAILED DESCRIPTION:
The application of PD-1/PD-L1 antibodies in cervical cancer is becoming increasingly widespread. However, monotherapy with PD-1 inhibitors demonstrates only a 10-20% response rate and a median progression-free survival of merely 2 months in patients with recurrent or metastatic cervical cancer. To address the issue of resistance to PD-1/PD-L1 antibodies in cervical cancer patients, we plan to conduct a clinical study. This study will administer a PD-1/CTLA-4 bispecific antibody to patients with recurrent or metastatic cervical cancer who are resistant to PD-1/PD-L1 therapy, thereby evaluating the efficacy and safety profile of the bispecific antibody in this specific patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent/metastatic cervical cancer who previously experienced failure of PD-1 blockade therapy;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
3. Life expectancy ≥3 months;
4. At least one measurable lesion per RECIST v1.1:

   Non-lymph node lesion: Longest diameter ≥10 mm Lymph node lesion: Short-axis diameter ≥15 mm Note: Previously irradiated lesions must be outside radiation fields or demonstrate progression post-radiation.
5. Adequate organ function within 14 days prior to treatment:

   1. Absolute neutrophil count (ANC) ≥1.0×10⁹/L
   2. Hemoglobin ≥60 g/L
   3. Platelet count ≥50×10⁹/L
   4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3×ULN (≤5×ULN for hepatic metastasis)
   5. Serum creatinine ≤2×ULN
6. Reproductive requirements:

   1. Non-childbearing potential (surgically sterilized or postmenopausal) OR
   2. Women of childbearing potential:

   Negative serum pregnancy test within 7 days prior to enrollment Commitment to use double-barrier contraception throughout the study and for 180 days post-treatment
7. Ability to comply with scheduled visits, treatment plans, and laboratory tests;
8. Voluntarily signed written informed consent.

Exclusion Criteria:

1. Prior treatment with anti-PD-1/CTLA-4 bispecific antibodies;
2. Active autoimmune disease requiring systemic control with corticosteroids (≥10 mg/day prednisone equivalent) or immunosuppressants within 14 days prior to enrollment;
3. Clinically significant cardiovascular/cerebrovascular events within 6 months prior to treatment, including:

   1. Acute myocardial infarction
   2. Unstable angina
   3. Cerebrovascular accident
   4. Symptomatic arterial/venous thrombosis or ischemic cardiomyopathy
   5. Clinically significant ventricular arrhythmias (sustained VT, VF, torsades de pointes)
   6. NYHA Class III/IV heart failure
   7. QTcF ≥480 ms or congenital long QT syndrome
   8. LVEF <50% or severe wall motion abnormality per echocardiography
   9. Uncontrolled hypertension (SBP >160 mmHg or DBP >100 mmHg)
   10. Other clinically significant arrhythmias (e.g., third-degree AV block);
4. Uncontrolled comorbidities potentially affecting protocol compliance:

   * Severe respiratory diseases (ILD, severe asthma)
   * Active infections:

     * HBV (HBsAg+ AND HBV-DNA >500 IU/mL)
     * HCV (HCV-Ab+ AND HCV-RNA+)
     * HIV-Ab+
     * Active TB or systemic infections requiring treatment ≤14 days
   * GI perforation/fistula ≤6 months (exceptions: resolved surgically)
   * Clinically significant bleeding ≤1 month (hematemesis, hemoptysis, etc.)
   * Active diverticulitis, abdominal abscess, or bowel obstruction;
5. Other malignancies within 3 years (excluding cured BCC, superficial bladder Ca, DCIS, or papillary thyroid Ca);
6. Known immunodeficiency disorders;
7. History of allogeneic hematopoietic stem cell or solid organ transplantation (excluding corneal grafts);
8. Systemic infections requiring IV antibiotics >7 days within 2 weeks prior to treatment;
9. Administration of live attenuated vaccines within 4 weeks before/after treatment;
10. Pregnancy or lactation;
11. Investigator-assessed ineligibility;
12. Concurrent participation in other clinical trials.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 1-year
  The objective response rate (ORR) assessed by the Independent Review Committee (IRC) (according to RECIST v1.1).

SECONDARY OUTCOMES:
DOR | 1-year
  The duration of response (DOR) assessed according to RECIST v1.1.
DCR | 1-year
  The disease control rate (DCR) assessed according to RECIST v1.1
OS | 1-year
  Time from diagnosis of disease to death due to any cause
PFS | 1-year
  Time from diagnosis of disease to disease progression or death due to any cause
Profile of adverse events | 3 years
  Frequency and severity of treatment-related toxicities, whether immune-related or non-immune-related

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Yuan, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital

IPD SHARING:
Plan to Share IPD: No